CLINICAL TRIAL: NCT07100340
Title: Feasibility and Safety of the Augmented Reality Guidance Software TAVIPILOT Software During Transcatheter Aortic Valve Replacement (TAVR/TAVI)
Acronym: SAITO 1B
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caranx Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 55003
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: TAVI(Transcatheter Aortic Valve Implantation)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TAVR procedure with TAVIPILOT Software (investigational medical device) (Experimental): Use of the TAVIPILOT Software during the procedure
  Interventions: Device: TAVR using a guidance software

INTERVENTIONS:
Device: TAVR using a guidance software — TAVR procedure with TAVIPILOT augmented reality guidance software operating during the procedure, enabling clinicians to assess the live analysis and recommendations provided by the software.

SUMMARY:
The TAVIPILOT Software by Caranx Medical is an advanced intraoperative assistance tool designed to enhance the accuracy of transcatheter aortic valve positioning during TAVI. It works alongside conventional fluoroscopy, using real-time image analysis to provide precise anatomical landmarks. TAVIPILOT Software detects key anatomical structures, tracks valve positioning, and uses AI-based confidence indicators to assist in alignment. The software is compatible with approved C-arm imaging systems and specific catheter models.

The objective is to assess the feasibility and safety of the TAVIPILOT Software augmented reality guidance software during TAVI procedures, aiming to improve valve positioning precision and, implicitly and to reduce implantation depth variations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥65
2. Indicated for transfemoral TAVR for severe aortic stenosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Investigational device-related safety | periprocedural
  The primary objective is to evaluate investigational device-related safety, including the occurrence of investigational device-related conversion to open-heart surgery, investigational device-related valve embolization.
Investigational device-related safety | Periprocedural
  The investigational device-related safety will also be assessed by verifying the absence of major technical malfunctions.

SECONDARY OUTCOMES:
Device usability | Periprocedural
  Evaluate clinical usability, assessed through customized questionnaires measuring clinician satisfaction, perceived ease of use, and integration of the devices into the procedural workflow.

IPD SHARING:
Plan to Share IPD: No